CLINICAL TRIAL: NCT03636269
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Intravenous CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus, With a 52-Week Open Label Extension
Brief Title: CR845-CLIN3103: A Global Study to Evaluate the Safety and Efficacy of CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus
Acronym: KALM-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR845-CLIN3103
Record Dates: First submitted 2018-08-03; First posted 2018-08-17 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Uremic Pruritus
Keywords: Hemodialysis; difelikefalin; CR845; Pruritus; Chronic Itch; Itch; Itching; Uremic Pruritus; Dialysis; CKD; CKD-associated pruritus; CKD-aP; ESRD (end stage renal disease); KALM; Chronic Kidney Disease; Kidney failure, chronic; Kidney dysfunction; Generalized pruritus
MeSH Terms: conditions — Pruritus; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — difelikefalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CR845 0.5mcg/kg (Active Comparator): IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
  Interventions: Drug: CR845 0.5 mcg/kg
- Placebo (Placebo Comparator): IV Placebo administered after each dialysis session (3 times/week)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR845 0.5 mcg/kg — IV CR845 0.5 mcg/kg administered three times/week
  Other Names: CR845; Difelikefalin
  Arms: CR845 0.5mcg/kg
Drug: Placebo — IV placebo administered three times/week
  Arms: Placebo

SUMMARY:
This is a multicenter, international study to evaluate the safety and efficacy of intravenous (IV) CR845 at a dose of 0.5 mcg/kg administered after each dialysis session. The study includes a 12-week randomized, double-blind, placebo-controlled Phase and a 52-week Open-label Extension Phase.

DETAILED DESCRIPTION:
Double-blind Phase: The Double-blind Phase of the study will consist of a Screening Visit, a 7-day Run-in Period, and a 12-week Double-blind Treatment Period. Informed consent will be obtained prior to performing any study-specific procedures. The Screening Visit will occur within 7 to 28 days prior to randomization to assess eligibility.

Open-label Extension Phase: Patients who received at least 30 doses of study drug (either active or placebo) during the 12-week Double-blind Treatment Period and continue to meet other eligibility criteria will have the option to receive open label CR845 for an additional 52 weeks.

The last dose of open-label study drug will be administered at the last dialysis visit on Week 52, or Early Termination.

Follow-up Period: A final safety Follow up Visit will be conducted 7-10 days after the End of Treatment/Early Termination Visit.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the Double-blind Phase of the study, a patient must meet the following criteria:

* Has end-stage renal disease (ESRD) and has been on hemodialysis 3 times per week for at least 3 months prior to the start of screening;
* Has at least 2 single-pool Kt/V measurements ≥1.2, or at least 2 urea reduction ratio measurements ≥65%, or 1 single pool Kt/V measurement ≥1.2 and 1 urea reduction ratio measurement ≥65% on different dialysis days during the 3 months period prior to screening;
* Prior to randomization:

  * Has completed Worst Itching Intensity NRS worksheets up to 8 days prior to 1st dose;
  * Has a mean baseline Worst Itching Intensity NRS indicative of moderate to severe uremic pruritus.
* To be eligible for inclusion into the Open-label Extension Phase of the study, each patient will have to fulfill the additional key following criteria at the time of entry into the Open-label Extension Phase:

  * Has received at least 30 doses of the planned 36 doses of study drug during the Double-blind Phase of this study;
  * Continues to meet inclusion criteria.

Key Exclusion Criteria:

A patient will be excluded from the Double-blind Phase of the study if any of the following criteria are met:

* Known noncompliance with dialysis treatment that in the opinion of the investigator would impede completion or validity of the study;
* Scheduled to receive a kidney transplant during the study;
* New or change of treatment received for itch including antihistamines and corticosteroids (oral, IV, or topical) within 14 days prior to screening;
* Received another investigational drug within 30 days prior to the start of screening or is planning to participate in another clinical study while enrolled in this study;
* Has pruritus only during the dialysis session (by patient report);
* Is receiving ongoing ultraviolet B and anticipates receiving such treatment during the study;
* Participated in a previous clinical study with CR845.
* A patient will be excluded from the Open-label Extension Phase of the study if any of the additional key following criteria are met at the time of entry into the Open-label Extension Phase:

  * Completed the Double-blind Phase of this study but exhibited adverse events during the course of the Treatment Period that may preclude continued exposure to the study drug;
  * Was noncompliant with protocol procedures during the Double-blind Phase of this study which is indicative of an inability to follow protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (92):
- United States (29):
  - Cara Therapeutics Study Site, Chula Vista, California
  - Cara Therapeutics Study Site, Fountain Valley, California
  - Cara Therapeutics Study Site, Northridge, California
  - Cara Therapeutics Study Site, Riverside, California
  - Cara Therapeutics Study Site 2, San Dimas, California
  - Cara Therapeutics Study Site, San Dimas, California
  - Cara Therapeutics Study Site, Westminster, Colorado
  - Cara Therapeutics Study Site, Hialeah, Florida
  - Cara Therapeutics Study Site, Miami Gardens, Florida
  - Cara Therapeutics Study Site, Orlando, Florida
  - Cara Therapeutics Study Site, Athens, Georgia
  - Cara Therapeutics Study Site, Macon, Georgia
  - Cara Therapeutics Study Site, Baton Rouge, Louisiana
  - Cara Therapeutics Study Site, Brockton, Massachusetts
  - Cara Therapeutics Study Site, Kalamazoo, Michigan
  - Cara Therapeutics Study Site, Roseville, Michigan
  - Cara Therapeutics Study Site, Saint Clair, Michigan
  - Cara Therapeutics Study Site, Tupelo, Mississippi
  - Cara Therapeutics Study Site, St Louis, Missouri
  - Cara Therapeutics Study Site, Clifton, New Jersey
  - Cara Therapeutics Study Site, Somerville, New Jersey
  - Cara Therapeutics Study Site, Albuquerque, New Mexico
  - Cara Therapeutics Study Site, Long Island City, New York
  - Cara Therapeutics Study Site, Austin, Texas
  - Cara Therapeutics Study Site, Dallas, Texas
  - Cara Therapeutics Study Site, McAllen, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, St. George, Utah
  - Cara Therapeutics Study Site, Roanoke, Virginia
- Australia (9):
  - Cara Therapeutics Study Site, Camperdown, New South Wales
  - Cara Therapeutics Study Site, Concord, New South Wales
  - Cara Therapeutics Study Site, Wahroonga, New South Wales
  - Cara Therapeutics Study Site, Westmead, New South Wales
  - Cara Therapeutics Study Site, Launceston, Tasmania
  - Cara Therapeutics Study Site, Clayton, Victoria
  - Cara Therapeutics Study Site, Heidelberg, Victoria
  - Cara Therapeutics Study Site, St Albans, Victoria
  - Cara Therapeutics Study Site, Adelaide
- Canada (5):
  - Cara Therapeutics Study Site, Halifax, Nova Scotia
  - Cara Therapeutics Study Site, Oshawa, Ontario
  - Cara Therapeutics Study Site, Scarborough Village, Ontario
  - Cara Therapeutics Study Site, Toronto, Ontario
  - Cara Therapeutics Study Site, Montreal, Quebec
- Czechia (2):
  - Cara Therapeutics Study Site, Frýdek-Místek
  - Cara Therapeutics Study Site, Prague
- Germany (2):
  - Cara Therapeutics Study Site, Düsseldorf
  - Cara Therapeutics Study Site, Heilbronn
- Hungary (7):
  - Cara Therapeutics Study Site, Baja
  - Cara Therapeutics Study Site, Debrecen
  - Cara Therapeutics Study Site 2, Pécs
  - Cara Therapeutics Study Site, Pécs
  - Cara Therapeutics Study Site, Szeged
  - Cara Therapeutics Study Site, Székesfehérvár
  - Cara Therapeutics Study Site, Szigetvár
- New Zealand (3):
  - Cara Therapeutics Study Site, Auckland
  - Cara Therapeutics Study Site, Hamilton
  - Cara Therapeutics Study Site, New Plymouth
- Poland (16):
  - Cara Therapeutics Study Site, Brodnica
  - Cara Therapeutics Study Site, Brzeg
  - Cara Therapeutics Study Site, Bydgoszcz
  - Cara Therapeutics Study Site, Grójec
  - Cara Therapeutics Study Site, Krakow
  - Cara Therapeutics Study Site, Kwidzyn
  - Cara Therapeutics Study Site 2, Lodz
  - Cara Therapeutics Study Site, Lodz
  - Cara Therapeutics Study Site, Nakło nad Notecią
  - Cara Therapeutics Study Site, Olkusz
  - Cara Therapeutics Study Site, Olsztyn
  - Cara Therapeutics Study Site, Poznan
  - Cara Therapeutics Study Site, Warsaw
  - Cara Therapeutics Study Site, Wroclaw
  - Cara Therapeutics Study Site, Zamość
  - Cara Therapeutics Study Site, Żyrardów
- South Korea (9):
  - Cara Therapeutics Study Site, Daegu
  - Cara Therapeutics Study Site 2, Daegu
  - Cara Therapeutics Study Site, Daejeon
  - Cara Therapeutics Study Site, Goyang-si
  - Cara Therapeutics Study Site, Guri-si
  - Cara Therapeutics Study Site, Seogu
  - Cara Therapeutics Study Site 2, Seoul
  - Cara Therapeutics Study Site 3, Seoul
  - Cara Therapeutics Study Site, Seoul
- Taiwan (4):
  - Cara Therapeutics Study Site, Kaohsiung City
  - Cara Therapeutics Study Site, New Taipei City
  - Cara Therapeutics Study Site 2, Taipei
  - Cara Therapeutics Study Site, Taipei
- United Kingdom (6):
  - Cara Therapeutics Study Site, Belfast
  - Cara Therapeutics Study Site, Ipswich
  - Cara Therapeutics Study Site, London
  - Cara Therapeutics Study Site, Londonderry
  - Cara Therapeutics Study Site, Nottingham
  - Cara Therapeutics Study Site, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fishbane SN, Block GA, Evenepoel P, Budden J, Morin I, Menzaghi F, Wen W, Lerma EV. Pruritus Severity and Serum Phosphate in CKD: A Post Hoc Analysis of Difelikefalin Studies. Kidney360. 2024 Sep 1;5(9):1270-1280. doi: 10.34067/KID.0000000000000520. Epub 2024 Jul 22. PMID 39037824
- [Derived] Weiner DE, Schaufler T, McCafferty K, Kalantar-Zadeh K, Germain M, Ruessmann D, Morin I, Menzaghi F, Wen W, Stander S. Difelikefalin improves itch-related sleep disruption in patients undergoing haemodialysis. Nephrol Dial Transplant. 2024 Jun 28;39(7):1125-1137. doi: 10.1093/ndt/gfad245. PMID 37968132
- [Derived] Fishbane S, Wen W, Munera C, Lin R, Bagal S, McCafferty K, Menzaghi F, Goncalves J. Safety and Tolerability of Difelikefalin for the Treatment of Moderate to Severe Pruritus in Hemodialysis Patients: Pooled Analysis From the Phase 3 Clinical Trial Program. Kidney Med. 2022 Jun 28;4(8):100513. doi: 10.1016/j.xkme.2022.100513. eCollection 2022 Aug. PMID 36039153
- [Derived] Topf J, Wooldridge T, McCafferty K, Schomig M, Csiky B, Zwiech R, Wen W, Bhaduri S, Munera C, Lin R, Jebara A, Cirulli J, Menzaghi F. Efficacy of Difelikefalin for the Treatment of Moderate to Severe Pruritus in Hemodialysis Patients: Pooled Analysis of KALM-1 and KALM-2 Phase 3 Studies. Kidney Med. 2022 Jun 28;4(8):100512. doi: 10.1016/j.xkme.2022.100512. eCollection 2022 Aug. PMID 36016762
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The ITT Population consisted of 473 subjects randomized to study treatment, 237 to difelikefalin and 236 to placebo. The Double-blind Safety Population consisted of 471 randomized subjects who received at least 1 dose of double-blind study drug during the Double-blind Treatment Period; 235 of these subjects were treated with difelikefalin, and 236 were treated with placebo. Two subjects were randomized to difelikefalin but did not receive any study drug.
Groups:
- Double-blind CR845 0.5mcg/kg; Open-label CR845 0.5mcg/kg: IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
  CR845 0.5 mcg/kg: IV CR845 0.5 mcg/kg administered three times/week
- Double-blind Placebo: IV Placebo administered after each dialysis session (3 times/week)
  Placebo: IV placebo administered three times/week
Period: Period 1: Double-blind Phase
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Open-label CR845 0.5mcg/kg
Started | 235 | 236 | 0
Completed | 206 | 223 | 0
Not Completed | 29 | 13 | 0
Not completed — Adverse Event | 13 | 7 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Eligibility (inclusion/exclusion criteria) | 2 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Other | 6 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Subject non-compliance | 1 | 2 | 0
Period: Period 2: Open-label Phase
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Open-label CR845 0.5mcg/kg
Started | 0 | 0 | 399
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 394
Not completed — Adverse Event | 0 | 0 | 21
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Eligibility (inclusion/exclusion criteria) | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 11
Not completed — Administrative | 0 | 0 | 36
Not completed — Other | 0 | 0 | 9
Not completed — Sponsor stopping study | 0 | 0 | 313

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Total
Number analyzed (Participants) | 235 | 236 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (13.11) | 59.6 (13.07) | 59.6 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 97 | 197
  Male | 135 | 139 | 274
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 12 | 20 | 32
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 53 | 38 | 91
  White | 162 | 169 | 331
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Itch Intensity as Assessed by the Percentage of Patients Achieving an Improvement From Baseline ≥3 Points With Respect to the Weekly Mean of the Daily 24-hour Worst Itching Intensity Numerical Rating Scale (NRS) Score at Week 12
Description: Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable". LS means estimated percent, odds ratio and P value used a logistic regression model.
Time Frame: Week 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CR845 0.5mcg/kg | Placebo
Number analyzed (Participants) | 237 | 236
percentage of subjects | 54.0 [43.9 to 63.9] | 42.2 [32.5 to 52.5]
Statistical Analysis 1: Comparison: CR845 0.5mcg/kg vs Placebo; Test type: Superiority; p = 0.020, Cui, Hung, Wang; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.08 to 2.41]

2. Secondary Outcome: Reduction of Itch Intensity as Assessed by the Percentage of Patients Achieving an Improvement From Baseline ≥4 Points With Respect to the Weekly Mean of the Daily 24-hour Worst Itching Intensity NRS Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo
Number analyzed (Participants) | 237 | 236
percentage of subjects | 41.2 [33.0 to 50.0] | 28.4 [21.3 to 36.7]
Statistical Analysis 1: Comparison: Double-blind CR845 0.5mcg/kg vs Double-blind Placebo; Test type: Superiority; p = 0.010, Cui, Hung, Wang; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.14 to 2.74]

3. Secondary Outcome: Improvement in Itch-related Quality of Life as Assessed by the Change From Baseline in Total Skindex-10 Scale Score at the End of Week 12
Description: The Skindex-10 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. The Skindex-10 has 10 questions; the total Skindex-10 score ranges from 0 to 60. A lower total score represents better quality of life.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo
Number analyzed (Participants) | 237 | 236
score on a scale | -16.6 [-19.3 to -14.0] | -14.8 [-17.4 to -12.2]
Statistical Analysis 1: Comparison: Double-blind CR845 0.5mcg/kg vs Double-blind Placebo; Test type: Superiority; p = 0.171, ANCOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.3 to 0.8], Standard Error of Mean 1.29

4. Secondary Outcome: Improvement in Itch-related Quality of Life as Assessed by the Change From Baseline in 5-D Itch Scale Score at the End of Week 12
Description: The 5-D Itch Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past 2 weeks. The questions cover five dimensions of itch including the degree, duration of itch/day, direction (improvement/worsening), disability (impact on activities such as work), and body distribution of itch. The 5-D Itch Scale has 5 questions; the total 5-D Itch Scale score ranges from 5 to 25, with higher scores indicating worse responses.
Time Frame: Baseline, Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo
Number analyzed (Participants) | 237 | 236
score on a scale | -4.9 [-5.6 to -4.2] | -3.8 [-4.5 to -3.1]
Statistical Analysis 1: Comparison: Double-blind CR845 0.5mcg/kg vs Double-blind Placebo; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.7 to -0.4], Standard Error of Mean 0.35

ADVERSE EVENTS:
Time Frame: The period of adverse event reporting will start after the signing of the informed consent form (ICF) through the study Follow-up Visit or Early Termination Visit (or 7 days after the last dose if no Early Termination Visit was conducted).
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Open-label CR845 0.5mcg/kg
All-Cause Mortality (participants affected / at risk) | 2/235 | 2/236 | 15/399
Serious Adverse Events (participants affected / at risk) | 58/235 | 51/236 | 130/399
Other Adverse Events (participants affected / at risk) | 56/235 | 43/236 | 204/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind CR845 0.5mcg/kg (N=235) | Double-blind Placebo (N=236) | Open-label CR845 0.5mcg/kg (N=399)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 6
Bradycardia (Cardiac disorders) | 2 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 5
Cardiac arrest (Cardiac disorders) | 1 | 1 | 3
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 3
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial ishaemia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 8 | 1 | 10
Pyrexia (General disorders) | 2 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 5
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pneumobilia (Hepatobiliary disorders) | 0 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 3 | 14
Cellulitis (Infections and infestations) | 2 | 1 | 1
Device related infection (Infections and infestations) | 2 | 1 | 4
Osteomyelitis (Infections and infestations) | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 3
Bronchitis (Infections and infestations) | 0 | 2 | 2
Influenza (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 22
Abscess limb (Infections and infestations) | 1 | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 3
Hepatic cyst infection (Infections and infestations) | 0 | 1 | 0
Incision site cellulitis (Infections and infestations) | 1 | 0 | 0
Infectious mononucloeosis (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 4
Skin infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 2
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Emphysematous cystitis (Infections and infestations) | 0 | 0 | 1
Gasteroenteritis (Infections and infestations) | 0 | 0 | 1
Gasteroenteritis escherichia coli (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 3 | 5
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 | 2 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0 | 6
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 3
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Chest x-ray abnormal (Investigations) | 0 | 1 | 0
Paracentesis (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2
Bleeding time prolonged (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 3 | 4
Fluid overload (Metabolism and nutrition disorders) | 0 | 2 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Delayed ischaemic neurological deficit (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1
Device malfunction (Product Issues) | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 3 | 0 | 5
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 3
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 7
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Abdominal hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Catheter placement (Surgical and medical procedures) | 0 | 0 | 1
Multiple drug therapy (Surgical and medical procedures) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 5 | 5
Peripheral ischaemia (Vascular disorders) | 3 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 3
Hypertensive crisis (Vascular disorders) | 0 | 2 | 3
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 1
Dry gangrene (Vascular disorders) | 0 | 0 | 2
Hypertensive emergency (Vascular disorders) | 0 | 0 | 2
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 1
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind CR845 0.5mcg/kg (N=235) | Double-blind Placebo (N=236) | Open-label CR845 0.5mcg/kg (N=399)
Diarrhoea (Gastrointestinal disorders) | 18 | 12 | 45
Vomiting (Gastrointestinal disorders) | 15 | 13 | 36
Fall (Injury, poisoning and procedural complications) | 14 | 11 | 52
Nausea (Gastrointestinal disorders) | 15 | 10 | 37
Dizziness (Nervous system disorders) | 12 | 12 | 31
Hypotension (Vascular disorders) | 9 | 4 | 25
Hypertension (Vascular disorders) | 6 | 10 | 24
Nasopharyngitis (Infections and infestations) | 3 | 5 | 22
Headache (Nervous system disorders) | 10 | 6 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 5 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03636269/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03636269/SAP_001.pdf